CLINICAL TRIAL: NCT02245347
Title: Genome Sequencing of MDR TB in Sputum
Brief Title: Genome Sequencing of Multidrug Resistant Tuberculosis (MDR TB) in Sputum
Acronym: MDRTB01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 12.LO.1694
Record Dates: First submitted 2014-09-12; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Tuberculosis
Keywords: TB; Tuberculosis; MDR TB; Drug resistant TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with expected MDR TB

SUMMARY:
Drug resistant tuberculosis is a growing problem world wide. The current methods for diagnosis are time consuming and may delay diagnosis and treatment for many weeks. In this study the investigators wish to take sputum samples from patients to see if the investigators can validate a molecular DNA based process for prompt identification of drug resistant tuberculosis. The investigators wish to extract and amplify DNA from drug resistant tuberculosis and identify genes within it that confer resistance.

DETAILED DESCRIPTION:
Drug resistant M. tuberculosis is an increasing problem in the United Kingdom and abroad. In the United Kingdom (UK) as a whole the number of isolates that were shown to be resistant to at least one of the first line drugs was nearly 400, with the total number of isolates approaching 5000. A total of 9040 cases were reported in the UK in 2009 and of these 6.9% demonstrated resistance to at least one first line drug(1). In certain populations the incidence of drug resistance is higher: in London, homeless patients, those who have been in prison and those from certain countries abroad, particularly Eastern Europe.

The difficulty of drug resistant tuberculosis is that the treatment duration, cost and complexity is increased. Typically the patient will be on treatment for 18 months or more and the Health Protection Agency (HPA) has estimated the cost of this as being upto £50000.

Current diagnosis rests on the culture of the M. tuberculosis and drug sensitivity testing. This can take six or eight weeks, meaning that patients may be on ineffective therapy for some time, leading to further transmission and deterioration of the patient's clinical condition. In this study the investigators would hope to develop a new test to improve and expedite the diagnosis of multi- drug resistant or MDR TB.

The predominant mechanism by which resistance occurs in M. tuberculosis is by the development and selection of mutants containing single nucleotide polymorphisms (SNP's)(2). Present commercial assays enable only a common subset (5-10) of the (900+) documented resistance mutations to be detected (www.tbdreamdb.com). It is highly likely that many more exist particularly in regions of the genome that may modulate sensitivity or resistance. This complexity is compounded by the requirement to treat TB with cocktails of antibiotics even for fully drug sensitive M.tuberculosis for which treatment consists of isoniazid (H), rifampicin (R), pyrazinamide (Z) and ethambutol (E). Multidrug resistant (MDR) and extensively drug resistant (XDR) TB cases are treated with second line drugs such as moxifloxacin, amikacin, capreomycin, para-aminosalicylic acid (PAS), thiocetazone and others for which genotypic markers of resistance are not tested. Such complex treatment combinations increase the need to screen multiple gene targets with the imperative to treat immediately with correct combinations of antibiotics.

The large number of mutations makes exhaustive detection of all known SNP's impossible with existing diagnostic procedures. Whole genome sequencing offers the potential to interrogate the genome of clinical isolates of M. tuberculosis for all known mutations and from this to infer an antimicrobial sensitivity pattern.

The extensive cost of treating and managing MDR cases(3) could potentially be reduced by obtaining a rapid genomic resistance profile early within the patients treatment. Cost benefit analysis of immediate whole genome sequencing (WGS) on all TB cases would be highly beneficial financially as well as clinically. The investigators propose to conduct a limited pilot study to assess the potential to acquire whole genome sequence directly from sputum specimens, early in a patient's treatment and to retrospectively define the potential impact of the availability of this data on patient care. This proposal will thus provide an evidence base for WGS to be developed into a routine diagnostic test/process with medical potential both at local National Health Service (NHS) level and globally so as to improve care pathways for MDR and XDR TB.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with smear positive tuberculosis who is capable to give informed consent will be offered to be included in the trial.

Exclusion Criteria:

* Any patient under 18 or who is unable to give informed consent will be excluded from this trial. Any patient who is unable to give a sputum sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smear positive patients with confirmed or suspected TB
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Identification and sequencing of mycobacterial DNA from sputum samples | within 24 hours of sample collection
  To see if mycobacterial DNA can be identified and sequenced from sputum and if the results correlate with the Microtiter Plate Methods done phenotypically in the standard manner.

CONTACTS AND LOCATIONS:
Locations (1):
- St George's NHS Healthcare Trust, London, United Kingdom